CLINICAL TRIAL: NCT02601235
Title: Clinical Evaluation of Safety and Efficacy of Pediatric Naridrin in Comparison to Afrin on the Improval of Nasal Congestion.
Brief Title: Efficacy and Safety of Pediatric Drugs in Nasal Congestion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMDEMS0214NA-III
Record Dates: First submitted 2015-11-05; First posted 2015-11-10 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Nasal Congestion
Keywords: nasal congestion
MeSH Terms: conditions — Nasal Obstruction | interventions — Naphazoline; Pyrilamine; dexpanthenol; Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naridrin (Experimental): Naridrin: 2 drops in each nostril once daily as prescription
  Interventions: Drug: Naridrin
- 0.05 % Oxymetazoline Hydrochloride (Active Comparator): 2 pumps in each nostril every 12 hours
  Interventions: Drug: Afrin

INTERVENTIONS:
Drug: Naridrin — Naridrin® : 2 drops in each nostril once daily as prescription
  Other Names: Naphazoline Hydrochloride; Mepyramine Maleate; Dexpanthenol
  Arms: Naridrin
Drug: Afrin — 2 pumps in each nostril every 12 hours.
  Other Names: oxymetazoline hydrochloride
  Arms: 0.05 % Oxymetazoline Hydrochloride

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Naridrin in improving nasal congestion.

DETAILED DESCRIPTION:
Open label, randomized, multicenter clinical study. Maximal experiment duration: 2 days; 2 visits. Safety and efficacy evaluation

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 10-17 years old with clinical symptoms of inflammatory of allergic nasal congestion in at least one nostril due to rhinitis or rhinopharyngitis (cold or flu);
* Signed Consent;
* Participants whose mother, father and / or legal guardian is in accordance with all study purposes and procedures;
* Participants with clinical symptoms of nasal congestion in at least one nostril diagnosed through the Glatzel mirror;
* Participants with minimal score of 2 points in the 0 to 3 scale (Moderate obstruction).

Exclusion Criteria:

* Participation in clinical trial in the year prior to this study;
* Total obstruction of one of the nostrils by other etiologies that are not inflammatory or allergic;
* Infectious bacterial-disease (clinically diagnosed);
* Participants treated with antibiotic or possible antibiotic use due to another medical condition;
* Use of intranasal corticosteroids (7 days prior to the study) or systemic (15 days prior to the study), regarding the plasma half-life of the drug;
* Use of decongestants or antihistamine (intranasal or systemic) in the 03 days prior to the study;
* Use of inhaled drugs (except nasal moisturizers such as saline solution) or treatment with immunosuppressants in the week before the study;
* Participants with septum deviation grade II and III, nasal polyps, severe turbinate hypertrophy, adenoid hypertrophy, or other determining factors for nasal obstruction;
* History of hyperthyroidism or hypertension;
* History of hypersensitivity to the components of the study drugs;
* History of transphenoidal hypophysectomy or oronasal surgery with exposure of the dura-mater;
* Exclusive mouth-breathers patients;
* Participants in chronic drug treatment for allergies (eg vaccines for allergy, cromolyn);
* History of alcohol and / or drug abuse 3 months prior to the study;
* Smokers
* Pregnancy or risk of pregnancy and lactating patients;
* PAny clinical, laboratory that, in the judgment of the investigator, may interfere with the safety of research participants.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 292 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Relief of Nasal Congestion | 2 days
  Relief of nasal congestion will be measured on a scale of 0 to 3 (0 = without congestion and 3 total congestion)

SECONDARY OUTCOMES:
Adverse Events | 2 days
  Safety of the drug will be assessed by observation of adverse events monitored for the type, frequency and intensity during the days of the follow-up.
  The evaluation of the heart frequency will also be a safety parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil